CLINICAL TRIAL: NCT02700542
Title: Asthma and Pest Control Study: Demonstrating Return-on-Investment for In-Home Pest Control for Children With Persistent Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York City Department of Health and Mental Hygiene (Other Government)
Collaborators: Montefiore Medical Center (Other); Healthfirst (Other); Affinity Health Plan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 13-097
Record Dates: First submitted 2015-03-31; First posted 2016-03-07 (Estimated); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Asthma
Keywords: asthma; pest management
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Active Comparator): Participants randomly assigned to the intervention group will receive the Integrated Pest Management (IPM) treatment 2-4 weeks of completion of the baseline assessment.The IPM protocol for this research will focus on pest control in the bathrooms and kitchen and will include an assessment of the pest problem, thorough cleaning, patching of small holes, identification and referral of any necessary large repairs, and targeted application of safe pesticides as needed. In cases of severe infestation, a second treatment visit might be required in the home.
  In addition to the intervention, the family will be provided with basic information about good pest-control practices, such as appropriate food storage, and be given a set of food storage containers.
  Interventions: Other: Integrated Pest Management
- Control (Placebo Comparator): Participants randomly assigned to the control group will be offered the equivalent intervention, information, and food storage containers after completion of their 12-month assessment.
  Interventions: Other: Integrated Pest Management

INTERVENTIONS:
Other: Integrated Pest Management — One-time, in-home, pest intervention for children with persistent asthma living in homes with parent-reported cockroach and/or mouse infestation.

SUMMARY:
The New York City Department of Health and Mental Hygiene and Montefiore Medical Center, with the Fund for Public Health of New York (FPHNY), DOHMH's fiscal agent, are partnering on a study to evaluate the feasibility, health outcomes and return-on-investment of a single, integrated pest management (IPM) intervention for Bronx, Harlem, and Northern Manhattan children aged 5 to 12 with persistent asthma who are living in homes with pests. By demonstrating cost effectiveness, this study could provide the basis for health insurance coverage of an IPM visit embedded in clinical treatment plans for high-risk asthma patients living with pests.

Asthma is the most common childhood disease in New York City, and both prevalence and hospitalization rates are highest in high-poverty neighborhoods. The greatest individual and community-level factor associated with asthma disparities is varying exposure to triggers in the home, most notably cockroaches and mice. Asthma health care costs are significant, and prevention efforts to reduce triggers could result in improved outcomes and significant cost savings. Unlike traditional pest control, which relies on pesticides, IPM eliminates pests and prevents re-infestation by addressing housing conditions conducive to pests and with safe, targeted use of pesticides. This project targets low-income children with the potential to significantly improve their health and well-being. A total of 400 families - 400+ children which includes screened and recruited siblings - will be recruited on to the study.

The study is designed to evaluate an inexpensive and scalable environmental intervention for asthma that can be replicated in other New York City neighborhoods and incorporated into any urban healthcare setting in New York State and nationwide.

DETAILED DESCRIPTION:
The New York City Department of Health and Mental Hygiene (DOHMH) and Montefiore Medical Center, with the Fund for Public Health of New York, DOHMH's fiscal agent, have partnered on a study to evaluate the feasibility, health outcomes and return-on-investment of a single integrated pest management (IPM) intervention for Bronx, Harlem and Northern Manhattan children aged 5 to 12 with persistent asthma who are living in homes with pests. Principal Investigator (PI) Daniel Kass, MSPH, Deputy Commissioner of the DOHMH Division of Environmental Health, has extensive experience overseeing evaluation of program and policy initiatives, and co-PI Marina Reznik, MD, MS, Associate Professor of Pediatrics at Montefiore, has conducted research on evaluating the impact of a home-based asthma intervention on asthma-related outcomes in children with persistent asthma recruited from Montefiore clinics.

Asthma is the most common childhood disease in New York City, and both prevalence and hospitalization rates are highest in high-poverty neighborhoods. The greatest individual and community-level factor associated with asthma disparities is varying exposure to triggers in the home, most notably cockroaches and mice. Asthma health care costs are significant, and prevention efforts to reduce triggers could result in improved outcomes and significant cost savings. Unlike traditional pest control, which relies solely on pesticides, IPM eliminates pests and prevents re-infestation by addressing housing conditions conducive to pests and with safe, targeted use of pesticides.

The specific goals of the project are to:

* Demonstrate the feasibility of implementing a basic IPM intervention in the homes of children aged 5-12 years with persistent asthma or current prescription for controller medication and past-year history of asthma-related urgent care visits living in households with pest problems.
* Evaluate changes in asthma outcomes and asthma-related health system utilization associated with the IPM intervention.
* Assess the costs and return-on-investment (ROI) for the IPM intervention.
* Report findings and support policies to adopt insurance reimbursement for basic IPM interventions embedded in health service delivery to prevent asthma exacerbations due to pest triggers in the home.

HealthFirst and Affinity, among the largest insurers of pediatric patients in the Bronx, are collaborating with the research team, providing support in recruitment and use of their data on health outcomes among study participants for the evaluation. The research team is also working with pest control experts to establish a well-priced and replicable protocol for IPM best practice. The protocol will build upon DOHMH's prior work to evaluate IPM in public housing, which demonstrated significant reductions in pest populations and allergens in kitchens and bedrooms, with sustained effects. The study aims to contribute to a best-practice model for one-time IPM service in the home that is not only effective in reducing asthma triggers but also practical and readily adoptable in the pest control industry, replacing the current pesticides-only approach. This groundwork is critical to efforts to scale up to meet demand, should IPM intervention become a reimbursable service in asthma care for high-risk children.

This two-year research project will employ a prospective, randomized controlled study design with the random assignment of 400 participants to two groups: intervention and control. Participants in both groups will be followed for a 12-month period with three assessments: at baseline (when recruited), 6 months, and 12 months after-recruitment. The intervention group will receive the IPM service within 2-4 weeks of completion of the baseline assessment. In addition to the intervention, the family will be provided with basic information about good pest-control practices, such as appropriate food storage, and be given a set of food storage containers. The control group will be provided basic pest control information at baseline and will be offered the equivalent intervention, information, and food storage containers after completion of their 12-month assessment. The primary clinical outcome measures will be: asthma-related urgent care (unscheduled ambulatory) visits, asthma-related emergency department (ED) visits, and asthma-related hospitalizations.

The evaluation of this proposed initiative will assess the intervention implementation and costs, its impact on health outcomes, healthcare cost savings or ROI.

This project targets low-income children with the potential to significantly improve their health and well-being. The study has been designed to evaluate an inexpensive and scalable environmental intervention for asthma that can be replicated in other New York City neighborhoods and incorporated into any urban healthcare setting in New York State and nationwide. By demonstrating cost effectiveness, this study could provide the basis for health insurance coverage of an IPM visit embedded in clinical treatment plans for high-risk asthma patients living with pests.

ELIGIBILITY:
Inclusion Criteria:

1. Current residence in the Bronx, Harlem and Northern Manhattan with no plans to move within the recruitment period (3 months) outside the Bronx, Harlem or Northern Manhattan

   a. Families with plans to move within the recruitment period to another location in the Bronx, Harlem, or Northern Manhattan will be placed on list to be called at the end of the recruitment period to reassess eligibility at that time, if the sample size has not yet been achieved.
2. Age: 5-12 years
3. Persistent asthma or currently prescribed inhaled corticosteroids/other prevention medication

   Persistent asthma (including mild, moderate or severe), according to National Heart Lung and Blood Institute (NHLBI) criteria:

   i. Experiencing symptoms more than 2 days per week in past month ii. Awaking at night due to symptoms more than 2 times per month iii. Use of SABA meds (i.e., albuterol) for symptom control (not prevention) more than 2 days per week in past month iv. Any interference with daily activity v. Having exacerbations requiring oral systemic corticosteroids 2 or more time per year
4. Any past-year urgent care visits for asthma:

   1. ED visits
   2. Hospitalizations
5. Parent-reported pest infestation - cockroaches or mice - in the home
6. Have a working phone
7. Caregiver primary language of English or Spanish

Exclusion Criteria:

1. Child living in foster care
2. Current residence in shelter or other similar temporary accommodation in the Bronx, Harlem, or Northern Manhattan

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 384 (Actual)
Dates: Start 2014-05-21 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in counts of urgent care (unscheduled ambulatory) visits at 6 months | Baseline to 6-months
Change from baseline in costs of urgent care (unscheduled ambulatory) visits at 6 months | Baseline to 6-Months
Change from 6-months in counts of urgent care (unscheduled ambulatory) visits at 12 months | 6 months and 12 months
Change from 6-months in costs of urgent care (unscheduled ambulatory) visits at 12 months | 6 months and 12 months
Change from baseline in counts of urgent care (unscheduled ambulatory) visits at 12 months | Baseline and 12 months
Change from baseline in costs urgent care (unscheduled ambulatory) visits at 12 months | Baseline and 12 months
Change from baseline in counts of Emergency Department visits at 6 months | Baseline to 6 months
Change from baseline in costs of Emergency Department visits at 6 months | Baseline to 6 months
Change from 6-months in counts of Emergency Department visits at 12 months | 6 month to 12 month
Change from 6-months in costs of Emergency Department visits at 12 months | 6 month to 12 month
Change from baseline in counts of Emergency Department visits at 12 months | Baseline to 12 months
Change from baseline in costs of Emergency Department visits at 12 months | Baseline to 12 months
Change from baseline in counts of hospitalizations at 6 months | Baseline to 6 months
Change from baseline in costs of hospitalizations at 6 months | Baseline to 6 months
Change from 6 months in counts of hospitalizations at 12 months | 6 months to 12 months
Change from 6 months in costs of hospitalizations at 12 months | 6 months to 12 months
Change from baseline in counts of hospitalizations at 12 months | Baseline to 12 months
Change from baseline in costs of hospitalizations at 12 months | Baseline to 12 months

SECONDARY OUTCOMES:
Change from baseline in number of symptom days per 2-weeks (Participant Reported Outcome) at 6 months | Baseline to 6 months
  Mean number of caregiver-reported asthma symptom days in the past 2 weeks (as per National Cooperative Inner-City Asthma Study), calculated as the maximum of 3 measures:
  i. Number of days when the child had wheezing, tightness in the chest, or cough; ii. Number of nights when the child lost sleep because of asthma iii. Number of days the child slowed down or stopped regular play or activities because of asthma.
Change from 6 months in number of symptom days per 2-weeks (participant Reported Outcome) at 12 months | 6 months to 12 months
  Mean number of caregiver-reported asthma symptom days in the past 2 weeks (as per National Cooperative Inner-City Asthma Study), calculated as the maximum of 3 measures:
  i. Number of days when the child had wheezing, tightness in the chest, or cough; ii. Number of nights when the child lost sleep because of asthma iii. Number of days the child slowed down or stopped regular play or activities because of asthma.
Change from baseline in number of symptom days per 2-weeks (participant reported outcome) at 12 months | Baseline to 12 months
  Mean number of caregiver-reported asthma symptom days in the past 2 weeks (as per National Cooperative Inner-City Asthma Study), calculated as the maximum of 3 measures:
  i. Number of days when the child had wheezing, tightness in the chest, or cough; ii. Number of nights when the child lost sleep because of asthma iii. Number of days the child slowed down or stopped regular play or activities because of asthma.
Change from Baseline in the Number of Days Child Missed School (Participant Reported Outcome) at 6 months | Baseline to 6 months
Change from 6 Months in the Number of Days Child Missed School (Participant Reported Outcome) at 12 months | 6 months to 12 months
Change from Baseline in the Number of Days Child Missed School (Participant Reported Outcome) at 12 months | Baseline to 12 months
Change from Baseline in the Number of Days Parent Missed Work (Participant Reported Outcome) at 6 Months | Baseline to 6 Months
Change from 6 Months in the Number of Days Parent Missed Work (Participant Reported Outcome) at 12Months | 6 Months to 12 Months
Change from Baseline in the Number of Days Parent Missed Work (Participant Reported Outcome) at 12Months | Baseline to 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Kass, MSPH, Principal Investigator — NYC Department of Health and Mental Hygiene; Marina Reznik, MD, MS, Principal Investigator — Montefiore Medical Center
Locations (2):
- United States (2):
  - New York City Department of Health and Mental Hygiene, New York, New York
  - Montefiore Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No